CLINICAL TRIAL: NCT02182024
Title: Pharmacokinetics, Pharmacodynamics, Safety and Tolerability of 150 mg Dabigatran Etexilate p.o. in Patients With Different Degrees of Renal Impairment in Comparison to Subjects With Normal Renal Function in a Monocentric, Open, Parallel-group Trial
Brief Title: Pharmacokinetics, Pharmacodynamics, Safety and Tolerability of Dabigatran Etexilate in Patients With and Without Renal Impairment
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1160.23
Record Dates: First submitted 2014-07-02; First posted 2014-07-08 (Estimated); Last update posted 2014-07-18 (Estimated); Status verified 2014-07

CONDITIONS: Renal Insufficiency
MeSH Terms: conditions — Renal Insufficiency | interventions — Dabigatran

ARMS (5):
- Dabigatran high dose in healthy subjects (Experimental): healthy subjects with a creatinine clearance of >80 mL/m
  Interventions: Drug: Dabigatran etexilate high dose
- Dabigatran high dose in mild renal impairment (Experimental): patients with a creatinine clearance of >50 up to 80 mL/min
  Interventions: Drug: Dabigatran etexilate high dose
- Dabigatran high dose in moderate renal impairment (Experimental): patients with a creatinine clearance of >30 up to 50 mL/min
  Interventions: Drug: Dabigatran etexilate high dose
- Dabigatran high dose in severe renal impairment (Experimental): patients with a creatinine clearance of up to 30 mL/min
  Interventions: Drug: Dabigatran etexilate high dose
- Dabigatran low dose in haemodialysis patients (Experimental): patients requiring haemodialysis
  Interventions: Drug: Dabigatran etexilate low dose

INTERVENTIONS:
Drug: Dabigatran etexilate high dose
  Arms: Dabigatran high dose in healthy subjects; Dabigatran high dose in mild renal impairment; Dabigatran high dose in moderate renal impairment; Dabigatran high dose in severe renal impairment
Drug: Dabigatran etexilate low dose
  Arms: Dabigatran low dose in haemodialysis patients

SUMMARY:
To assess the effect of different degrees of renal impairment on the pharmacokinetics and pharmacodynamics of dabigatran etexilate administered orally.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male or female subjects determined by results of screening with a creatinine clearance >80 mL/min (group 1, control group)
* Renally impaired male or female subjects determined by results of screening with the following creatinine clearance results:

  * creatinine clearance >50 - ≤80 mL/min (group 2)
  * creatinine clearance >30 - ≤50 mL/min (group 3)
  * creatinine clearance ≤30 mL/min (group 4)
  * uraemia requiring maintenance dialysis (group 5)
  * Signed written informed consent in accordance with Good Clinical Practice (GCP) and local legislation
* Age >=18 and <=75 years
* BMI >=18.0 and <=32 kg/m2, at least 45 kg for females

Exclusion Criteria:

* Any finding of the medical examination (including blood pressure, pulse rate, and electrocardiogram) deviating from normal and of clinical relevance
* Clinically relevant gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunologic or hormonal disorders
* Surgery of gastrointestinal tract (except appendectomy, cholecystectomy or herniotomy)
* Clinically relevant diseases of the central nervous system
* Relevant history of orthostatic hypotension, fainting spells or blackouts
* Abnormal prothrombin time (PT), TT, aPTT (must be within the normal range after no more than one repeated test), thrombocytes <150000/μl (two repeats of the first test)
* Evidence of haematuria either macroscopically detectable or microscopic on urinalysis (normal microscopic results after no more than one repeated test)
* Evidence of blood dyscrasia, haemorrhagic diathesis, severe thrombocytopenia, cerebrovascular haemorrhage, bleeding tendencies associated with active ulceration or overt bleeding of gastrointestinal, respiratory or genitourinary tract or any disease or condition with haemorrhagic tendencies (e.g. cerebral aneurysm, dissecting aorta, central nervous system (CNS) trauma, retinopathy or nephrolithiasis)
* Recent or contemplated diagnostic or therapeutic procedures with potential for uncontrollable bleeding (e.g. spinal puncture, lumbar block anaesthesia, surgery of CNS or eye or surgery resulting in large open surfaces) within 14 days before or after drug administration of this clinical trial
* Chronic or relevant acute infections
* History of allergy/hypersensitivity (including drug allergy) which is deemed relevant to the trial as judged by the investigator
* For women with childbearing potential: no reliable contraception (accepted methods are intra uterine device, hormonal contraceptives, bilateral tubal ligation, hysterectomy, condoms) or pregnancy (known or detected by a positive pregnancy test) or breast feeding period
* Intake of drugs with a long half-life (>24 hours) (<1 month prior to administration or during the trial)
* Use of any drugs, within 14 days prior to administration or during the trial
* Participation in another trial with an investigational drug (<2 months prior to drug administration or during trial)
* Drug abuse
* Blood donation or loss >400 mL, <1 month prior to administration or during the trial
* Excessive physical activities <5 days prior to administration of study drug or during trial
* Clinically relevant laboratory abnormalities

Renally impaired subjects (groups 2, 3, 4 and 5) who met any of the following criteria were not be entered into this trial:

* Moderate and severe concurrent liver function impairment (e.g. due to hepatorenal syndrome)
* Clinically relevant gastrointestinal, respiratory, cardiovascular, metabolic, immunologic or hormonal disorders
* Surgery of gastrointestinal tract (except appendectomy, cholecystectomy or herniotomy)
* Clinically relevant diseases of the central nervous system
* Relevant history of orthostatic hypotension, fainting spells or blackouts
* Abnormal values for PT, TT, aPTT and thrombocytes considered by the investigator or one of the co-investigators to be clinically relevant
* Evidence of blood dyscrasia, haemorrhagic diathesis, severe thrombocytopenia, cerebrovascular haemorrhage, bleeding tendencies associated with active ulceration or overt bleeding of gastrointestinal, respiratory or genitourinary tract or any disease or condition with haemorrhagic tendencies (e.g. cerebral aneurysm, dissecting aorta, CNS trauma, retinopathy, nephrolithiasis) considered by the investigator or one of the co-investigators to be clinically relevant
* Recent or contemplated diagnostic or therapeutic procedures with potential for uncontrollable bleeding (e.g. spinal puncture, lumbar block anaesthesia, surgery of CNS or eye or surgery resulting in large open surfaces) within 14 days before or after drug administration of this clinical trial
* Chronic or relevant acute infections
* History of allergy/hypersensitivity (including drug allergy) which is deemed relevant to the trial as judged by the investigator
* For women with childbearing potential: no reliable contraception (accepted methods are intra-uterine device, hormonal contraceptives, bilateral tubal ligation, hysterectomy or condoms) or pregnancy (known or detected by a positive pregnancy test) or breast-feeding period
* Participation in another trial with an investigational drug (<2 months prior to administration or during trial)
* Drug abuse
* Blood donation or loss >400 mL, <1 month prior to administration or during the trial
* Excessive physical activities < 5 days prior to administration of study drug or during trial
* Clinically relevant laboratory abnormalities except those values typical for renally impaired patients

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2005-04; Primary Completion 2006-03 (Actual)

PRIMARY OUTCOMES:
AUC0-infinity (area under the concentration time curve of the analyte in plasma over the time interval from 0 extrapolated to infinity) | pre-dose and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 48 and 72 h after administration, additional 96 h in subjects with severe renal impairment and dialysis patients
Cmax (maximum concentration of the analyte in plasma) | pre-dose and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 48 and 72 h after administration, additional 96 h in subjects with severe renal impairment and dialysis patients
CL/F (apparent clearance of the analyte in the plasma after extravascular administration) | pre-dose and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 48 and 72 h after administration, additional 96 h in subjects with severe renal impairment and dialysis patients
international normalized ratio (INR) | pre-dose and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 48 and 72 h after administration, additional 96 h in subjects with severe renal impairment and dialysis patients
activated partial thromboplastin time (aPTT) | pre-dose and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 48 and 72 h after administration, additional 96 h in subjects with severe renal impairment and dialysis patients
Ecarin clotting time (ECT) | pre-dose and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 48 and 72 h after administration, additional 96 h in subjects with severe renal impairment and dialysis patients
thrombin time (TT) | pre-dose and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 48 and 72 h after administration, additional 96 h in subjects with severe renal impairment and dialysis patients

SECONDARY OUTCOMES:
AUC0-tz (area under the concentration-time curve of the analyte in plasma over the time interval from 0 to the time of the last quantifiable data point) | pre-dose and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 48 and 72 h after administration, additional 96 h in subjects with severe renal impairment and dialysis patients
AUCt1-t2 (area under the concentration-time curve of the analyte in plasma over the time interval t1 to t2, time interval to be determined) | pre-dose and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 48 and 72 h after administration, additional 96 h in subjects with severe renal impairment and dialysis patients
tmax (time from dosing to the maximum concentration of the analyte in plasma, oral administration only) | pre-dose and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 48 and 72 h after administration, additional 96 h in subjects with severe renal impairment and dialysis patients
λz (terminal rate constant in plasma) | pre-dose and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 48 and 72 h after administration, additional 96 h in subjects with severe renal impairment and dialysis patients
t1/2 (terminal half-life of the analyte in plasma) | pre-dose and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 48 and 72 h after administration, additional 96 h in subjects with severe renal impairment and dialysis patients
MRTpo (mean residence time of the analyte in the body after p.o. administration) | pre-dose and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 48 and 72 h after administration, additional 96 h in subjects with severe renal impairment and dialysis patients
Vz/F (apparent volume of distribution during the terminal phase λz following an extravascular dose) | pre-dose and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 48 and 72 h after administration, additional 96 h in subjects with severe renal impairment and dialysis patients
Ae0-72 (amount of analyte that is eliminated in urine from the time interval 0 to 72 h) | pre-dose over 12 hours and post dose in fractions of 0 - 12, 12 - 24, 24 - 48, and 48-72 h, additional until 96 h in subjects with severe renal impairment
fe0-72 (fraction of administered drug excreted unchanged in urine from time point 0 to 72 h) | pre-dose over 12 hours and post dose in fractions of 0 - 12, 12 - 24, 24 - 48, and 48-72 h, additional until 96 h in subjects with severe renal impairment
CLR,0-72 (renal clearance of the analyte in plasma from the time point 0 h until the timepoint 72 h) | pre-dose over 12 hours and post dose in fractions of 0 - 12, 12 - 24, 24 - 48, and 48-72 h, additional until 96 h in subjects with severe renal impairment
Plasma protein binding of dabigatran | within 1 h before study drug administration
Changes from baseline in pulse rate | Day 4, Day 5 in patients with renal impairment
Changes from baseline in systolic and diastolic blood pressure | Day 4, Day 5 in patients with renal impairment
Changes from baseline in ECG | Day 4, Day 5 in patients with renal impairment
Changes from baseline in routine laboratory | Day 4, Day 5 in patients with renal impairment
Occurrence of adverse events | up to day 4, up to day 5 in patients with renal impairment
Assessment of tolerability on a 4-point scale | Day 4, Day 5 in patients with renal impairment